CLINICAL TRIAL: NCT05139121
Title: A Phase 3, Multicenter, Open-Label, Single Arm Study of MR-100A-01 in Women of Childbearing Potential to Evaluate Contraceptive Efficacy and Safety
Brief Title: Study of the Safety and Efficacy of MR-100A-01 in Approximately 1200 Healthy Women for up to 13 Cycles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Technologies Inc. (Industry)
Collaborators: Mylan Inc. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MR-100A-01-TD-3001
Record Dates: First submitted 2021-10-20; First posted 2021-12-01 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Contraception
Keywords: Birth Control; Pregnancy Prevention; Contraceptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MR-100A-01 (Experimental): MR-100A-01 is a transdermal delivery system designed to deliver daily hormone exposure of Norelgestromin and Ethinyl Estradiol
  Interventions: Drug: MR-100A-01

INTERVENTIONS:
Drug: MR-100A-01 — Transdermal contraceptive delivery system
  Other Names: Transdermal contraceptive delivery system

SUMMARY:
Study of the contraceptive efficacy, cycle control, safety, and tolerability of MR-100A-01 in approxmiately 1200 women for up to 13 cycles

DETAILED DESCRIPTION:
MR-100A-01 is a TDS of norelgestromin 4.86 mg/ethinyl estradiol 0.264 mg. This study will evaluate the contraceptive efficacy, cycle control, safety, and tolerability of MR-100A-01.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, post-menarcheal and premenopausal women at risk of pregnancy who are at least 16 years of age with no upper age limit. Post-menarcheal female subjects who are at risk of pregnancy, and <18 years are eligible provided that:

   1. Applicable national, state, and local laws allow the subject to consent to sexual intercourse,
   2. Applicable national, state, and local laws allow subjects in this age group to consent/assent to receive contraceptive services, and
   3. All applicable laws and regulations regarding the informed consent/assent of the subjects to participate in clinical trials are observed.
2. Desires to avoid pregnancy, is seeking to use hormonal contraception for at least 1 year.
3. Has negative UPT results at screening and at enrollment visits.
4. Has normal, regular menstrual cycles that are between 21 and 35 days.
5. Engages in regular heterosexual vaginal intercourse.
6. Agrees not to use other contraceptives or other methodology to prevent pregnancy during the study.
7. Able to understand and voluntarily provide written informed consent or assent to participate in the study.
8. Able to understand and willing to be compliant with study procedures.
9. Willing to accept a risk of pregnancy.
10. Has demonstrated ability to complete e-Diary.
11. Planning to reside within a reasonable driving/ public transport distance of the research site (approximately 150 miles) for around 12 months (13 cycles).

Exclusion Criteria:

1. Known or suspected pregnancy or planning pregnancy during next 12 months.
2. Subjects with known hypersensitivity or intolerance to estrogens, progestins, or any components of the MR-100A-01 product.
3. History or presence of dermal sensitivity to topical applications including bandages, surgical tape.
4. Known infertility (current or known history) or history of sterilization in either partner.
5. Received injectable hormonal contraceptive therapy within 10 months of study enrollment or has had less than 2 consecutive, spontaneous menses after an injectable hormonal contraceptive was received at least 10 months earlier.
6. Current use of hormonal contraceptive implants (still implanted; or if an implant was removed, less than 3 consecutive spontaneous menses have occurred between removal and enrollment).
7. Has non-hormonal or hormonal intrauterine device (IUD) in place or has had a recent IUD removal without one spontaneous menses after removal prior to the date of enrollment.
8. Recent surgical or medical abortion, miscarriage, ectopic pregnancy, or vaginal or cesarean delivery and have had less than 3 consecutive, spontaneous menses or withdrawal bleeding episodes prior to enrollment.
9. Subjects lactating at the time of screening into the study.
10. Anticipates routine use of condoms or any other form of back-up contraception for protection from sexually transmitted infections during the study or for emergency contraception.
11. Subjects having a known contraindication to combined hormonal contraception as listed below:

    1. Smoker who is ≥35 years old.
    2. History or presence of ischemic heart disease, coronary artery disease, myocardial infarction, stroke, other cerebrovascular diseases including transient ischemic attacks (TIAs), valvular heart disease with complications (pulmonary hypertension, risk for atrial fibrillation, or history of subacute bacterial endocarditis), peripartum cardiomyopathy.
    3. History or presence of hypertension (including adequately controlled hypertension) or hypertension with vascular disease or elevated blood pressure (BP) defined as systolic BP ≥140 mm Hg or diastolic BP ≥90 mm Hg, measured in sitting position after 5 minutes of rest, considering the average of two readings measured 1 to 2 minutes apart
    4. History or presence of deep vein thrombosis/pulmonary embolism (DVT/PE) or superficial venous thrombosis.
    5. Has any comorbid condition that may require major surgery with prolonged immobilization during the study period.
    6. Subjects with known inherited or acquired hypercoagulopathy.
    7. History or presence of systemic lupus erythematosus.
    8. History or presence of neurological conditions including migraine with aura at any age, migraine without aura in women ≥35 years age or in women who smoke, or multiple sclerosis with prolonged immobility.
    9. History or presence of or suspected carcinoma of breast.
    10. Has diabetes mellitus with nephropathy, retinopathy, neuropathy, or other vascular disease or diabetes of >20 years' duration.
    11. Has inflammatory bowel disease (ulcerative colitis or Crohn's disease) who are at increased risk for VTE
    12. Medically treated or presence of symptomatic gall bladder disease.
    13. History of combined hormonal contraceptive/pregnancy-related cholestasis/jaundice.
    14. Presence of liver disease.
    15. History of organ transplantation within 5 years before screening or chronic disease potentially necessitating organ transplantation during the anticipated course of the study.
    16. Subject has requirement to be on treatment with medications prohibited during study.
12. Known or suspected estrogen or progestin sensitive malignant or premalignant conditions.
13. History of any other condition that in the Investigator's opinion suggests an elevated risk of arterial or venous thromboembolic disease.
14. Has uncontrolled thyroid disorder.
15. Has diagnosis of hereditary angioedema.
16. Has hyperlipidemia on screening.
17. Has uncontrolled diabetes mellitus.
18. Subjects with abnormal significant liver function tests.
19. Has a significantly abnormal cervical cancer screening test (cervical cytology with reflex human-papilloma-virus (HPV) testing or with HPV co-testing) performed at screening visit (for subjects aged ≥21 years) i.e., cervical dysplasia or invasive cervical cancer or has any abnormal cytology with/without HPV testing during 6 months prior to screening which may require additional screening or treatment during the study period
20. Subjects with chlamydial or gonorrheal infection.
21. Has unexplained vaginal bleeding.
22. History of known or suspected hepatitis B or C infection or high risk for sexually transmitted disease (STD).
23. Known human immunodeficiency virus (HIV) infection or positive confirmatory test at screening.
24. Current known active infection of coronavirus disease 2019 (COVID-19) or increased risk of COVID-19 related morbidity. Subjects who have had previous COVID-19 infections but have recovered by the time of enrollment visit may be enrolled if there are no current COVID-19 symptoms; Subjects who had previously received COVID-19 vaccine may be enrolled irrespective of the timing of the vaccination.
25. Within the past year, either history of suicidal ideation or attempt or severe depression requiring hospitalization.
26. Presence of any other concomitant disease or laboratory result that may worsen under hormonal treatment based on Investigator's discretion.
27. Positive urine drug screen.
28. Recent history (within prior 12 months) of drug or alcohol abuse or at Investigator discretion, history greater than 12 months prior and at risk for noncompliance. Current or recent history of (recreational or medicinal) marijuana use is not exclusionary at the investigator's discretion upon assessment of any potential risk.
29. Participation in an investigational study within 30 days prior to enrollment or intention to participate within next 13 months.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1319 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Contraceptive efficacy of MR-100A-01 when used over thirteen 28-day cycles in healthy, post-menarcheal, premenopausal, heterosexually active female subjects of childbearing potential who are at least 16 years of age and at risk of pregnancy | 12 months (13 cycles)
  The primary efficacy endpoint will be pregnancy rate described by Pearl Index (PI). PI is defined as the number of pregnancies per 100 women-years times 100

SECONDARY OUTCOMES:
Cycle-wise pregnancy rates over 1 year evaluated using life table analysis [secondary efficacy] | 12 months (13 cycles)
  The rate of cycle-wise pregnancies
Cumulative pregnancy rates over 1 year evaluated using life table analysis [secondary efficacy] | 12 months (13 cycles)
  The rate of cycle-wise pregnancies
Method failure Pearl Index (PI) [secondary efficacy] | 12 months (13 cycles)
  The method failure PI is defined as PI among all complete or incomplete on therapy cycles in which intercourse occurred and protocol guidelines were not followed
Incidence of adverse events (AEs) [safety and tolerability] | 12 months (13 cycles)
  The number of AEs
Incidence of serious adverse events (SAEs) [safety and tolerability] | 12 months (13 cycles)
  The number of SAEs
Incidence of application site reactions [safety and tolerability] | 12 months (13 cycles)
  The number of application site reactions
Number of episodes of scheduled and unscheduled bleeding [cycle control] | 12 months (13 cycles)
  The number of incidences of scheduled and unscheduled bleeding
Number of days of scheduled and unscheduled bleeding [cycle control] | 12 months (13 cycles)
  The observed number of days of scheduled or unscheduled bleeding
Proportion of subjects reporting scheduled and unscheduled bleeding [cycle control] | 12 months (13 cycles)
  The number of subjects reporting scheduled and unscheduled bleeding
Adhesion performance as measured by adhesion scores [patch adhesion] | 12 months (13 cycles)
  The descriptive figures of adhesion performance

CONTACTS AND LOCATIONS:
Locations (100):
- United States (96):
  - Mobile Ob-Gyn, P.C., Mobile, Alabama
  - Velocity Clinical Research, Mobile, Alabama
  - Mesa Obstetricians and Gynecologists., Mesa, Arizona
  - Precision Trials AZ, Phoenix, Arizona
  - Visions Clinical Research Tucson, Tucson, Arizona
  - Alliance Research Institute, Bell Gardens, California
  - Essential Access Health, Berkeley, California
  - Velocity Clinical Research - Huntington Park, Huntington Park, California
  - Essential Access Health, Los Angeles, California
  - Axis Clinical Trials, Los Angeles, California
  - Matrix Clinical Research, Los Angeles, California
  - Velocity Clinical Research - Gardena, Los Angeles, California
  - Velocity Clinical Research, Panorama City, Los Angeles, California
  - Stanford University, School of Medicine, Department of Obstetrics and Gynecology, Palo Alto, California
  - Empire Clinical Research, Pomona, California
  - Northern California Research Corp, Sacramento, California
  - Women's Health Care Research Corp., San Diego, California
  - Wr-McCr, Llc, San Diego, California
  - Amicis Research Center, San Fernando, California
  - Red Rocks Ob-Gyn, Lakewood, Colorado
  - IntimMedicine Specialists, Washington D.C., District of Columbia
  - Quantum Clinical Trials, Boynton Beach, Florida
  - Aventura OB/GYN Associates, Hallandale, Florida
  - CenExel RCA, Hollywood, Florida
  - Global Research Associates, Homestead, Florida
  - UF Health Woman's Specialist - Emerson, Jacksonville, Florida
  - Multi-Specialty Research Associates, Lake City, Florida
  - WR-Multi-Specialty Research Associates LLC, Lake City, Florida
  - Altus Research, Lake Worth, Florida
  - Ob-Gyn Associates Of Mid-Florida, PA, Leesburg, Florida
  - Advanced Pharma CR LLC, Miami, Florida
  - Avantis Clinical Research, Miami, Florida
  - AdMed Research, LLC, Miami, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - ProCare Research Center, Corp., Miami Gardens, Florida
  - Global Health Research Center, Miami Lakes, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Healthcare Clinical Data, Inc. - Segal Institute for Clinica, North Miami, Florida
  - Clintheory Healthcare Miami, Orlando, Florida
  - Physician Care Clinical Research, Sarasota, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Agile Clinical Research Trials, Atlanta, Georgia
  - Medisense Inc., Atlanta, Georgia
  - CenExel iResearch Atlanta, LLC, Decatur, Georgia
  - Soapstone Center for Clinical Research, Decatur, Georgia
  - WR-Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - CenExel iResearch, LLC, Savannah, Georgia
  - Fellows Research Alliance, Inc., Savannah, Georgia
  - Velocity Clinical Research, Boise, Meridian, Idaho
  - Clinical Trials Management, Covington, Louisiana
  - Velocity Clinical Research - Covington, Covington, Louisiana
  - Praetorian Pharmaceutical Research, LLC, Marrero, Louisiana
  - Velocity Clinical Research Metairie, Metairie, Louisiana
  - Javara Inc/Privia Medical Group, LLC, Chevy Chase, Maryland
  - SBL Special Services, Frederick, Maryland
  - Planned Parenthood of Minnesota, Minneapolis, Minnesota
  - Excel Clinical Research, Las Vegas, Nevada
  - Office of Edmond Pack, MD, Las Vegas, Nevada
  - Wake Research Clinical Research Center of Nevada - Emergency Medicine, Las Vegas, Nevada
  - Hassman Research Institute, Marlton, New Jersey
  - Velocity Clinical Research- Albuquerque, Albuquerque, New Mexico
  - Bosque Women's Care, Albuquerque, New Mexico
  - New York Clinical Trials - Brooklyn, Brooklyn, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - Javara Inc. Tryon Medical-South Park, Charlotte, North Carolina
  - Carolina Women's Research And Wellness Center, Durham, North Carolina
  - Unified Women's Clinical Research Raleigh, Raleigh, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Unified Women's Clinical Research d/b/a Lyndhurst Clinical R, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Velocity Clinical Research, Cleveland, Cleveland, Ohio
  - Aventiv Research - Columbus, Dublin, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Oregon Health & Science University Center for Women's Health, Portland, Oregon
  - Ob/Gyn Associates Of Erie, Erie, Pennsylvania
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Velocity Clinical Research-Charleston, Charleston, South Carolina
  - Venus Gynecology, LLC., Myrtle Beach, South Carolina
  - Chattanooga Medical Research LLC, Chattanooga, Tennessee
  - Alliance for Multispecialty Research, LLC., Knoxville, Tennessee
  - WR-Medical Research Center of Memphis, LLC., Memphis, Tennessee
  - DCT-HCWC, LLC dba Discovery Clinical Trials, Dallas, Texas
  - Cedar Health Research, Irving, Texas
  - Advances In Health, Inc., Pearland, Texas
  - Physicians' Research Options, LLC Corner Canyon Clinic, Draper, Utah
  - Physicians' Research Options, LLC, Pleasant Grove, Utah
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Velocity Clinical Research - Salt Lake City, West Jordan, Utah
  - Tidewater Clinical Research/TPW, Norfolk, Virginia
  - Eastern Virginia Medical School, Clinical Research Center, Norfolk, Virginia
  - Virginia Women's Health Associates, Reston, Virginia
  - Seattle Clinical Research Center, Seattle, Washington
- Canada (3):
  - Centricity Research Quebec City, Lévis, Quebec
  - Diex Recherche Victoriaville, Victoriaville, Quebec
  - Clinique RSF Inc., Québec
- Puerto Rico Medical Research, Inc, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: No